CLINICAL TRIAL: NCT04774328
Title: A Three-Part, Phase 1/2, Randomized, Double-blind, Placebo-Controlled, Adaptive Safety, Pharmacokinetics, and Preliminary Efficacy Study of CA-008 (Vocacapsaicin) in Patients Undergoing Ventral Hernia Repair
Brief Title: Preliminary Study of CA-008 (Vocacapsaicin) in Patients Undergoing Ventral Hernia Repair
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Concentric Analgesics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CA-PS-209
Record Dates: First submitted 2021-02-24; First posted 2021-03-01 (Actual); Results first posted 2022-09-14 (Actual); Last update posted 2022-09-14 (Actual); Status verified 2022-08

CONDITIONS: Postsurgical Pain
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- CA-008 (vocacapsaicin) (Active Comparator): Single administration
  Interventions: Drug: CA-008 (vocacapsaicin)
- Placebo (Placebo Comparator): Single administration
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: CA-008 (vocacapsaicin) — Single administration of CA-008 (vocacapsaicin) versus placebo
  Arms: CA-008 (vocacapsaicin)
Drug: Placebo — Single administration of CA-008 (vocacapsaicin) versus placebo
  Arms: Placebo

SUMMARY:
A Three-Part, Phase 1/2, Randomized, Double-blind, Placebo-Controlled, Adaptive Safety, Pharmacokinetics, and Preliminary Efficacy Study of CA-008 (Vocacapsaicin) in Patients Undergoing Ventral Hernia Repair

ELIGIBILITY:
Inclusion Criteria:

* Scheduled elective, primary, open laparotomy with VHR, with retromuscular, preperitoneal mesh placement, with midline fascial reconstruction
* ASA physical class 1, 2, or 3
* BMI </= 40 kg/m2
* Aged 18-80 years old

Exclusion Criteria:

* Concurrent condition requiring analgesic treatment during study period
* Opioid tolerant
* Known allergy to capsaicin or other study medication
* Use of prohibited medications

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2020-09-09 (Actual); Primary Completion 2021-06-15 (Actual); Study Completion 2021-06-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Daneshvari Solanki, MD, Principal Investigator — First Surgical Hospital
Locations (1):
- First Surgical Hospital, Houston, Texas, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The clinical trial was conducted at one clinical research surgical center from September 2020 until June 2021. Qualified patients are adults aged 18 to 80 years of age, inclusive, who are planning to undergo an elective, open laparotomy for ventral hernia repair (VHR), with retromuscular, preperitoneal mesh repair and who otherwise meet eligibility criteria.
Pre-assignment Details: Sixty-seven patients were screened. Ten met requirements for open-label Part A and 24 were randomized to Part B. Patients meeting all inclusion and no exclusion criteria underwent VHR surgery and dosing on Day 1. The patient was closely followed during the outpatient portion to Day 29 post surgery. Part A began enrolling in September 2020 and Part B on 10FEB2021.
  Part C was not conducted due to a corporate decision, and not due to any safety concerns.
Groups:
- CA-008 (Vocacapsaicin), 15 mg - Part A: Single administration of CA-008 (vocacapsaicin), 15 mg (50 ml of a 0.3 mg/mL solution)
  Open-label, feasibility and safety assessment, exploration of different delivery techniques
- CA-008 (Vocacapsaicin), 24 mg - Part B: CA-008 (vocacapsaicin): single administration of CA-008 (vocacapsaicin), 24 mg (80 ml of a 0.3 mg/mL solution)
  Double-blind, randomized, placebo-controlled, parallel-group design.
- Placebo - Part B: Single administration of placebo
  Double-blind, randomized, placebo-controlled, parallel-group design.
Period: Overall Study
Arm/Group | CA-008 (Vocacapsaicin), 15 mg - Part A | CA-008 (Vocacapsaicin), 24 mg - Part B | Placebo - Part B
Started | 10 | 12 | 12
Follow-up to 29 Days Post Surgery | 10 | 12 | 12
Completed | 10 | 12 | 12
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- CA-008 (Vocacapsaicin), 15 mg - Part A: Single administration of CA-008 (vocacapsaicin), 15 mg (50 ml of a 0.3 mg/mL solution)
- CA-008 (Vocacapsaicin), 24 mg - Part B: Single administration of CA-008 (vocacapsaicin), 24 mg (80 ml of a 0.3 mg/mL solution)
- Placebo - Part B: Single administration of placebo
- Total: Total of all reporting groups
Arm/Group | CA-008 (Vocacapsaicin), 15 mg - Part A | CA-008 (Vocacapsaicin), 24 mg - Part B | Placebo - Part B | Total
Number analyzed (Participants) | 10 | 12 | 12 | 34
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 10 | 12 | 12 | 34
  >=65 years | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 47.9 (10.8) | 47.1 (10.16) | 42.2 (10.19) | 45.6 (10.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 4 | 3 | 9
  Male | 8 | 8 | 9 | 25
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 8 | 6 | 15
  Not Hispanic or Latino | 9 | 4 | 6 | 19
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 1 | 0 | 1 | 2
  White | 9 | 12 | 11 | 32
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 10 | 12 | 12 | 34

OUTCOME MEASURES:

1. Primary Outcome: Pain at Rest - Part B
Description: Pain at rest measured by a Numeric Rating Scale (NRS) from time 0 to 96 hours (AUC 0-96). NRS pain scores at rest were collected at 1, 2, 4, 6, 8, 12, 16, 20, 24 and every 4 hours there after post the time of entry into the PACU (while the patient is awake), until discharge from the inpatient until at 96 hour. NRS area under the curve (AUC) is the weighted sum of current pain intensity assessments for a specified time interval. The NRS ranks pain from 0-10; zero being no pain present and 10 being the worst possible pain. Other than 0 and 10, no other pain ratings (2-9) were labeled.
Time Frame: Up to 96 hours
Population: modified Intent to Treat (mITT) population
Measure: Mean (Standard Deviation); unit: score on a scale*hours
Groups:
- CA-008 (Vocacapsaicin), 24 mg - Part B: Single administration of CA-008 (vocacapsaicin), at a fixed dose of 24 mg (80 mL of a 0.3 mg/mL concentration)
Arm/Group | CA-008 (Vocacapsaicin), 24 mg - Part B | Placebo - Part B
Number analyzed (Participants) | 12 | 12
score on a scale*hours | 148.98 (146.68) | 188.26 (120.60)
Statistical Analysis 1: Comparison: CA-008 (Vocacapsaicin), 24 mg - Part B vs Placebo - Part B; Test type: Other — Analysis of Variance (ANOVA); p = 0.4812, ANOVA; Median Difference (Final Values) = -39.28, 95% CI 2-sided [-152.97 to 74.40], Standard Error of Mean 54.818

2. Secondary Outcome: Evoked NRS - Part B
Description: Evoked NRS pain scores (three maneuvers: coughing, sitting up, walking) from time 0-96 hours. Evoked NRS scores were obtained twice daily in the morning at 10:00AM (± 1h) and in the afternoon at 4:00PM (±1 h).
  NRS area under the curve (AUC) is the weighted sum of current pain intensity assessments for a specified time interval. The NRS ranks pain from 0-10; zero being no pain present and 10 being the worst possible pain. Other than 0 and 10, no other pain ratings (2-9) were labeled.
Time Frame: Up to 96 hours
Population: modified Intent to Treat (mITT) population
Measure: Mean (Standard Deviation); unit: score on a scale*hours
Arm/Group | CA-008 (Vocacapsaicin), 24 mg - Part B | Placebo - Part B
Number analyzed (Participants) | 12 | 12
score on a scale*hours
  Coughing | 187.58 (176.49) | 345.66 (135.50)
  Sitting-up | 116.24 (105.90) | 171.28 (105.69)
  After ambulation | 143.42 (112.71) | 222.14 (94.89)
Statistical Analysis 1: Comparison: CA-008 (Vocacapsaicin), 24 mg - Part B vs Placebo - Part B; Applies to evoked measure of "after coughing"; Test type: Other — ANOVA; p = 0.0222, ANOVA; Mean Difference (Final Values) = -158.08, 95% CI 2-sided [-291.29 to -24.87], Standard Error of Mean 64.232
Statistical Analysis 2: Comparison: CA-008 (Vocacapsaicin), 24 mg - Part B vs Placebo - Part B; Applies to evoked measure for "after sitting up"; Test type: Other — ANOVA; p = 0.2158, ANOVA; Mean Difference (Final Values) = -55.04, 95% CI 2-sided [-144.61 to 34.53], Standard Error of Mean 43.190
Statistical Analysis 3: Comparison: CA-008 (Vocacapsaicin), 24 mg - Part B vs Placebo - Part B; Applies to evoked measure of "after ambulation"; Test type: Other — ANOVA; p = 0.0777, ANOVA; Mean Difference (Final Values) = -78.73, 95% CI 2-sided [-166.93 to 9.48], Standard Error of Mean 42.532

3. Secondary Outcome: Opioid Consumption - Part B
Description: Total opioid consumption (OC) converted to an oral morphine equivalent (OME) dose from 0 to 96 hours (OC 0-T96) and 0 to Day 8 (OC 0-D8).
Time Frame: Up to Day 8
Population: modified Intent to Treat (mITT) population
Measure: Mean (Standard Deviation); unit: mg morphine equivalents
Groups:
- CA-008 (Vocacapsaicin), 24 mg: Single administration of CA-008 (vocacapsaicin), at a fixed dose of 24 mg (80 mL of a 0.3 mg/mL concentration)
- Placebo: Single administration of Placebo
Arm/Group | CA-008 (Vocacapsaicin), 24 mg | Placebo
Number analyzed (Participants) | 12 | 12
mg morphine equivalents
  OC 0 to 96 hours | 27.18 (31.63) | 36.56 (30.70)
  OC 0 to Day 8 | 29.68 (37.66) | 37.81 (33.27)
Statistical Analysis 1: Comparison: CA-008 (Vocacapsaicin), 24 mg vs Placebo; Entry applies to OC 0-96 hours; Test type: Other — ANOVA; p = 0.4690, ANOVA; Mean Difference (Final Values) = -9.375, 95% CI 2-sided [-35.764 to 17.014], Standard Error of Mean 12.7245
Statistical Analysis 2: Comparison: CA-008 (Vocacapsaicin), 24 mg vs Placebo; Applies to OC 0 - Day 8; Test type: Other — ANOVA; p = 0.5811, ANOVA; Mean Difference (Final Values) = -8.125, 95% CI 2-sided [-38.208 to 21.958], Standard Error of Mean 14.5059

ADVERSE EVENTS:
Time Frame: All AEs were recorded through at least 29 days, and on average 30.8 days, after the completion of surgery.
Description: The definition of adverse events is consistent with clinicaltrials.gov definitions.
  Additional optional information: verbatim terms used by Investigators to identify AEs were coded by system organ class (SOC) and PT using the Medical Dictionary for Regulatory Activities (MedDRA Version 24.0).
Arm/Group | CA-008 (Vocacapsaicin), 15 mg - Part A | CA-008 (Vocacapsaicin), 24 mg - Part B | Placebo - Part B
All-Cause Mortality (participants affected / at risk) | 0/10 | 0/12 | 0/12
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/12 | 0/12
Other Adverse Events (participants affected / at risk) | 9/10 | 10/12 | 10/12
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | CA-008 (Vocacapsaicin), 15 mg - Part A (N=10) | CA-008 (Vocacapsaicin), 24 mg - Part B (N=12) | Placebo - Part B (N=12)
Bradycardia (Cardiac disorders) | 1 (1) | 1 (1) | 0 (0)
Tachycardia (Cardiac disorders) | 0 (0) | 3 (3) | 2 (2)
Abdominal discomfort (Gastrointestinal disorders) | 1 (1) | 1 (1) | 1 (1)
Abdominal distension (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Abdominal pain lower (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 6 (6) | 6 (6) | 8 (8)
Flatulence (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 2 (2) | 4 (4) | 1 (1)
Vomiting (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0)
Chest pain (General disorders) | 0 (0) | 1 (1) | 0 (0)
Discomfort (General disorders) | 0 (0) | 0 (0) | 1 (1)
Hypersensitivity (Immune system disorders) | 0 (0) | 1 (1) | 0 (0)
Postoperative wound infection (Infections and infestations) | 0 (0) | 0 (0) | 2 (2)
Incision site rash (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Incision site vesicles (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 2 (2)
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Blood Pressure Increased (Investigations) | 0 (0) | 1 (1) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Dizziness (Nervous system disorders) | 1 (1) | 2 (2) | 1 (1)
Headache (Nervous system disorders) | 2 (2) | 0 (0) | 0 (0)
Tachypenoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Blister (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 1 (1)
Hypertension (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Disclosure restriction on the PI and/or institution:

1. Sponsor can embargo communications or publications regarding trial results for more than 60 days but less than 181 days from the time submitted to the sponsor. The sponsor cannot extend the embargo.
2. The Institution and Investigator agree that any Institutional Publication shall be made after the Multicenter Publication, provided that the Multicenter Publication is submitted within eighteen (18) months after conclusion of the Study.

DOCUMENTS (2):
  • Study Protocol (2021-03-15): https://cdn.clinicaltrials.gov/large-docs/28/NCT04774328/Prot_000.pdf
  • Statistical Analysis Plan (2021-05-14): https://cdn.clinicaltrials.gov/large-docs/28/NCT04774328/SAP_001.pdf